CLINICAL TRIAL: NCT02270957
Title: Clarification of Abatacept Effects in SLE With Integrated Biologic and Clinical Approaches (The ABC Study)
Brief Title: Clarification of Abatacept Effects in SLE With Integrated Biologic and Clinical Approaches
Acronym: ABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMRF 13-38
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept (Active Comparator): Patients receive Abatacept 125 mg subcutaneously weekly for six months. An optional continuation up until 12 months is allowed. Background immune suppressants are withdrawn at the beginning of the study and the option of depomedrol up to 320 mg total (in divided doses) is allowed at any time up through the visit 2 months after study medication is started. After this additional rescue is allowed with any standard of care treatment and/or open label abatacept (since patients are blinded) but this additional rescue will define non-response in the primary endpoint at six months.
  Interventions: Biological: Abatacept
- Placebo (Placebo Comparator): Patients receive placebo instead of Abatacept in a double blind fashion. Otherwise participation is the same, including that at the time of treatment failure they may elect any standard of care treatment and/or to begin taking open label abatacept but this rescue will define non-response in the primary endpoint at six months.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Abatacept
  Other Names: Orencia
  Arms: Abatacept
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled trial of abatacept for the treatment of lupus arthritis and other manifestations of lupus. Patients with lupus and at least 3 tender and 3 swollen joints and </= 20 mg prednisone have other background immune suppressants withdrawn at entry. They can elect to receive up to a total of 320 mg depomedrol (in two or more injections) between the screening visit and the visit 2 months after dosing begins. Abatacept (125 mg) or placebo is administered in weekly subcutaneous doses. After 3 months of treatment patients who are not responding may elect to receive open label abatacept with or without additional standard of care therapies. Such patients are considered non responders. The primary endpoint is the British Isles Lupus Assessment Group Index (BILAG)-linked Combined Lupus Assessment (BICLA) which will require a clinically significant improvement in arthritis and other active features of lupus

DETAILED DESCRIPTION:
Research Hypothesis: Abatacept is effective in lupus arthritis and this will be discernible in a small trial with robust endpoints which incorporates withdrawal of background immune suppressants

Study Schematic: Abatacept 125 mg or placebo will be given in a 1:1 randomization subcutaneously each week for six months. All patients may elect to continue six more months on open label Abatacept. Background Immune Suppressants will be withdrawn at any time between screening and the first dosing visit. At or after screening, patients may elect 40-160 mg depomedrol shots prn not to exceed 320 mg total up to and including the Month 2 Visit (two months after the first dosing visit) After that, additional steroids or immune suppressants, if necessary, will be allowed but the patient will be considered a non-responder in the primary endpoint at six months on that basis. At of after the 3 month visit patients with significant clinical flare may also elect to receive open label Abatacept but will be considered non-responders in the primary endpoint at six months.

Primary Objective: To compare response rates between Abatacept-Treated and Placebo-Treated Patients with active lupus arthritis in a trial designed with background immune suppressant withdrawal, limited steroid rescue, and a robust, discriminatory endpoint. The trial design and primary endpoint of response by BICLA (defined below) have been pre-tested by us for safety and ability to ensure placebo group non-response, underscoring our powering of the study. This will support a rational decision about further development of abatacept for SLE at minimal cost.

Secondary clinical outcome measures used as endpoints will include: SRI 4/5, changes in joint counts, SLEDAI, BILAG, CLASI, PGA, and LFA REAL measures.

The definitions of the clinical outcome measures are as follows: BICLA: BILAG-based Combined Lupus Assessment, This is defined as British Isles Lupus Assessment Group (BILAG) index scores that were severe at entry (BILAG A scores) improving to a moderate (BILAG B) level (or better) and all features that were moderate at entry improving to a mild level (BILAG C scores) or resolved (BILAG D scores) without increase in any other BILAG feature or SLEDAI scoring (see SLEDAI definition below), as well as no more than 10% worsening in a Physician's Global Assessment or any additional treatments after the protocolized baseline rescue (e.g. no new SLE treatments after the two month visit). SLEDAI stands for the Systemic Lupus Erythematosis Disease Activity Index. SRI 4/5 is defined as SLEDAI improvement by at least 4 points (or 5 points respectively), no increase in BILAG-measured disease activity and no more than 10% worsening in a Physician's Global Assessment (PGA). CLASI stands for the Cutaneous Lupus Erythematosus Disease Area and Severity Index. PGA stands for Physician's Global Assessment. LFA REAL stands for the Lupus Foundation of America Rapid Evaluation of the Activity of Lupus. This instrument is in a pilot phase but will be tested in the ABC study.

PK and immunogenicity studies will also be performed to help in interpretation of outcomes. Novel biologic discovery will be integrated into the clinical trial to support both pre-specified and exploratory biomarker discovery. Data will be generated that might be used to help select more appropriate patient subsets for future trials and, along with PK data, help to guide optimal dosing strategies. Optimizing patient selection and dosing are important goals for further increasing demonstrable effect size in trials by increasing the response rates in the treatment group.

This study will be performed as a double blind, randomized, placebo-controlled clinical trial with 1:1 randomization of patients to abatacept 125 mg weekly subcutaneous dose or placebo, with the withdrawal of background immune suppressants. Limited steroid rescue is allowed between the screening visit and the Month 2 visit per protocol. Additional standard of care rescue medications may be used after that as needed but will define non-response at the primary endpoint date of six months. Flaring patients may elect to receive open label abatacept at Month 3 but will also be defined as non-responders in the primary endpoint. All patients may elect to receive open label abatacept for an additional six months after the primary endpoint date, with two follow up visits (2 and 4 months post medication withdrawal) to assess withdrawal effects and to complete the safety assessments.

Accrual Goal: This study will continue to recruit until we achieve the goal of 60 patients who complete study visits through the 6 month endpoint.

Correlative Studies: Extensive exploratory protocol-specific and ancillary immune pharmacodynamic studies, focusing first on changes in IFN alpha, BLyS and other B Cell pathways. A major focus will also be on T Cell pathways with a focus on T suppressor/TH17 dichotomy after treatment with abatacept. A responder analysis will be performed in order to generate hypotheses useful for selecting appropriate patients for this treatment and optimizing dosing strategies.

Adverse Events, Serious Adverse Events and Adverse Events of special interest (infusion reactions and infections) will be collected and described. Stopping Rules: Patients may be withdrawn by the investigator for non-compliance or safety. All patients terminating before six months will be considered non responders in the primary analysis. Use of off protocol immune suppressants will not necessarily dictate withdrawal but will determine non-responder status. A DSMB board of at least two physicians (four are currently participating) will review data and may stop the study if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Four 1997 revised ACR Classification Criteria for SLE
3. Active polyarticular arthritis meeting at minimum BILAG 2004 B definition with a minimum of 3 tender and 3 swollen joints observed at the screening visit
4. Men and women 18 to 70 years of age.
5. Women of childbearing potential and men with partners of childbearing potential must use an acceptable method of birth control throughout the study
6. Women of childbearing potential must have a negative urine pregnancy test at screening and Study Day 1 (baseline visit) and may not be breast feeding

Exclusion Criteria:

1. Current severe, organ-threatening disease (e.g. acute nephritis appropriate for induction therapy, CNS lupus (excepting chorea, cranial neuropathy, and resolving optic neuritis) or any lupus condition requiring cyclophosphamide, biologic therapy, or IV bolus steroids of >/= 500 mg.
2. Subjects who are incapable of understanding or completing study-related assessments.
3. Subjects with any condition, whether or not related to SLE, which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
4. Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ.
5. Subjects who currently abuse drugs or alcohol.
6. Subjects with acute herpes zoster or cytomegalovirus (CMV) within 2 months of screening.
7. Subjects who have received any live vaccines within 3 months of first dose.
8. Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
9. Subjects at risk for tuberculosis (TB).
10. Subjects known to be positive for hepatitis B surface antigen or hepatitis C unless negative by PCR or RIBA
11. Acute hemolytic anemia with hemoglobin < 7.0 g/dL or known change in Hg by 2.0 g/dL within four months
12. WBC < 2500/mm3 (< 3 x 109/L) unless due to chronic stable lupus activity
13. Platelets < 40,000/mm3 (< 3 x 109/L) (If less than 100,000 must have been stable (within a range of 10,000/mm3 ) within two months of screening or in two tests during the screening period.
14. Serum creatinine > 2 times the ULN
15. Serum ALT or AST > 2.5 times the ULN
16. Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
17. Known allergy/sensitivity to the study agent or carrier.
18. Treatment with investigational drug within 28 days (or 5 terminal half-lives) of the Day 1 dose.
19. Cyclophosphamide within 3 months of Day 1 or bolus IV steroids >/=500 mg within 1 month
20. Prednisone > 20 mg qd after the screening visit

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan T Merrill, MD, Study Director — Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified results through an application process, linked to our institutional research cohorts, where there is a standard operating procedure approval process where research is deemed to be appropriate and relevant to SLE
Supporting Information: Study Protocol
Time Frame: June 2021-May 2023
Access Criteria: contact the PI at joan-merrill@omrf.org

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Thanou A, James JA, Arriens C, Aberle T, Chakravarty E, Rawdon J, Stavrakis S, Merrill JT, Askanase A. Scoring systemic lupus erythematosus (SLE) disease activity with simple, rapid outcome measures. Lupus Sci Med. 2019 Dec 30;6(1):e000365. doi: 10.1136/lupus-2019-000365. eCollection 2019. PMID 31921432

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: Patients receive Abatacept 125 mg subcutaneously weekly for six months. An optional continuation up until 12 months is allowed. Background immune suppressants are withdrawn at the beginning of the study and the option of depomedrol up to 320 mg total (in divided doses) is allowed at any time up through the visit 2 months after study medication is started. After this additional rescue is allowed with any standard of care treatment and/or open label abatacept (since patients are blinded) but this additional rescue will define non-response in the primary endpoint at six months.
  Abatacept
- Placebo: Patients receive Placebo but at the time they meet non-response criteria they may elect open label abatacept or any standard of care to treat their SLE
Period: Overall Study
Arm/Group | Abatacept | Placebo
Started | 31 | 35
Completed | 27 | 31
Not Completed | 4 | 4
Not completed — Lack of Efficacy | 2 | 4
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients receive Placebo. At any time that they meet non-response criteria (primary endpoint) they may elect to be treated with any standard of care medication or open label abatacept Placebo
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.9) | 46.9 (11.9) | 45.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 26 | 43
  African | 8 | 6 | 14
  Asian | 0 | 0 | 0
  Native American/Alaskan Native | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 31 | 35 | 66
anti-dsDNA positive [Number; unit: participants] | 5 | 12 | 17
low complement [Number; unit: participants] | 5 | 9 | 14
Number with at least one BILAG "B" score [Count of Participants; unit: Participants] — The BILAG stands for British Isles Lupus Assessment Group. The BILAG Index is an outcome measure that uses a glossary and a set of scoring rules based on progress over the prior month, in order to assign disease activity in each of nine organ systems as "A" (severe), "B" (moderate) or "C" (mild activity) vs no active disease in prior month.
  Participants | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: British Isles Lupus Assessment Group Index-based Combined Lupus Assessment (BICLA)
Description: The British Isles Lupus Assessment Group Index is a scoring system for progress of disease activity over the prior month with a scoring system that rates each organ system as "A" or severe, "B" or moderate, "C" or mild vs no activity in the past month. To meet the BICLA endpoint requires all baseline severe features (BILAG A) improving to moderate (BILAG B), mild or resolved, and all baseline BILAG B features improving to mild or resolved without increase in any other feature on either the BILAG or a different measure called the SLEDAI (SLE Disease Activity Index). Furthermore there must be no increase in Physician's Global Assessment or any rescue medications after the month 2 visit. Only those meeting all of these criteria meet the primary endpoint.
Time Frame: 6 months
Population: Full Analysis Set: All Randomized Patients
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Patients receive Abatacept 125 mg subcutaneously weekly for six months. An optional continuation up until 12 months is allowed. Background immune suppressants are withdrawn at the beginning of the study and the option of depomedrol up to 320 mg total (in divided doses) is allowed at any time up through the visit 2 months after study medication is started. After this additional rescue is allowed with any standard of care treatment and/or open label abatacept (since patients are blinded) but this additional rescue will define non-response in the primary endpoint at six months.
  Placebo
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 31 | 35
Participants | 8 | 8
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p > 0.999, Chi-squared

2. Post Hoc Outcome: SLE Responder Index-4 (SRI-4)
Description: Comparing the endpoint date at six months to Baseline, there must be a 4 point decreased in SLEDAI score (SLEDAI is defined as the SLE Disease Activity Index). The SLEDAI is a discontinuous scale in which each type of sign or symptom of active SLE is assigned a fixed number of points. Although the scale includes possible signs or symptoms adding up to more than 100 points it is rare for any (even very severe) patient to ever have a total score > 20. To meet the SLE Responder Index endpoint, There must also be no worsening of BILAG (British Isles Lupus Assessment Group Index (described in the primary endpoint section) and no worsening of PGA (a visual analogue scale reflecting physicians global assessment) by more than 10% of the scale. To meet this endpoint there must also be no new or increased medication initiated after Baseline other than the steroid rescues up to Month 2.
Time Frame: 6 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Patients receive Placebo but if the primary endpoint is met as "non-response" at any time they may elect any standard of care treatment or may initiate abatacept open label.
  Placebo
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 31 | 35
Participants | 9 | 8
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.587, Chi-squared

3. Post Hoc Outcome: 4 Point Improvement in the SLE Disease Activity Index (SLEDAI)
Description: The SLEDAI is a discontinuous scoring system that weights disease activity not by severity of individual symptoms but by the weighting of organs. This makes it less robust for comparing one group of patients to another, but it is quite useful to gave numbers of patients with improvement, since to lower the score a rigorous improvement must be documented
Time Frame: Comparison of Baseline to 6 months
Population: Full Analysis Set of all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 31 | 35
Participants | 9 | 8
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.587, Chi-squared — None of the endpoints were met in any pre-specified unbiased Full Analysis Set analysis

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Abatacept: Patients receive Abatacept 125 mg subcutaneously weekly for six months.
- Placebo: Patients receive Placebo subcutaneously weekly for six months.
Arm/Group | Abatacept | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/31 | 4/35
Other Adverse Events (participants affected / at risk) | 29/31 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=31) | Placebo (N=35)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe gastroenteritis leading to hospitalization
viral syndrome (Infections and infestations) | 1 (1) | 1 (1) — viral sepsis
sickle cell crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — R tib/fib fracture
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
cardiac valve dysfunction (Cardiac disorders) | 0 (0) | 1 (1) — aortic and mitral valve dysfunction and replacement
opiate overdose (Social circumstances) | 0 (0) | 1 (1)
respiratory compromise (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — prolonged hospitalization from opiate overdose
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) — prolonged hospitalization after opiate overdose
blocked ureter (Renal and urinary disorders) | 0 (0) | 1 (1) — stent placement
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=31) | Placebo (N=35)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
gastroenteritis (Gastrointestinal disorders) | 17 (18) | 11 (11)
oral candida (Infections and infestations) | 0 (0) | 8 (8)
injection site reaction (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) — all mild or moderate and none led to discontinuation
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6) — these were not expected rashes due to SLE all were suspected drug reactions but all self limited and not leading to discontinuation
otitis media (Ear and labyrinth disorders) | 1 (1) | 4 (5)
urinary tract infection (Infections and infestations) | 5 (7) | 17 (24)
upper respiratory infection (Infections and infestations) | 15 (20) | 16 (27)
influenza (Infections and infestations) | 1 (1) | 3 (4)
sinusitis (Infections and infestations) | 4 (4) | 8 (14)
vaginal yeast infestation (Infections and infestations) | 1 (1) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02270957/Prot_SAP_000.pdf